CLINICAL TRIAL: NCT07265180
Title: Oxytocin-Augmented Mindfulness-Based Group Psychotherapy for Patients With Schizophrenia Spectrum Disorders - an Oxytocin-dose Comparison (OXYMIND2.0)
Brief Title: Oxytocin-Augmented Group Psychotherapy for Patients With Schizophrenia - an Oxytocin-dose Comparison
Acronym: OXYMIND2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Kerem Böge, Prof. Dr. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OXYMIND2.0
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Schizophrenia Spectrum Disorders (SSD)
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oxytocin (24 I.U. Syntocinon®) (Active Comparator): The patients received a spray of synthetic oxytocin (24 I.U. Syntocinon®) in combination with mindfulness-based group therapy (MBGT) over 4 weeks once a week. Due to an effect latency of 30-80 min after intranasal administration of oxytocin on social behavior, the dose was administered 30 min before the 50 min session.
  Interventions: Other: Oxytocin
- Oxytocin (48 I.U. Syntocinon®) (Active Comparator): The patients received a spray of synthetic oxytocin (48 I.U. Syntocinon®) in combination with mindfulness-based group therapy (MBGT) over 4 weeks once a week. Due to an effect latency of 30-80 min after intranasal administration of oxytocin on social behavior, the dose was administered 30 min before the 50 min session.
  Interventions: Other: Oxytocin
- Placebo (Placebo Comparator): The patients received a placebo nasal spray in combination with mindfulness-based group therapy (MBGT) over 4 weeks once a week. Due to an effect latency of 30-80 min after intranasal administration of oxytocin on social behavior, the dose was administered 30 min before the 50 min session.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Oxytocin — Oxytocin nasal spray in combination with mindfulness based group therapy (MBGT).
  Arms: Oxytocin (24 I.U. Syntocinon®); Oxytocin (48 I.U. Syntocinon®)
Other: Placebo — Placebo nasal spray in combination with mindfulness based group therapy (MBGT).
  Arms: Placebo

SUMMARY:
The effectiveness of current treatment options for sociocognitive deficits and negative symptoms (NS) in schizophrenia spectrum disorders (SSD) remains limited. The cause of NS is thought to be an interference between the mesocorticolimbic dopamine system for social reward expectancy and the network for socioemotional processes. Oxytocin (OXT) may enhance functional connectivity between these neuronal networks. Lower plasma OXT levels correlate negatively with NS severity and deficits in social cognition in SSD. It has been shown that intranasal OXT administration improves social cognition in healthy subjects but in SSD results are inconsistent. According to the social salience hypothesis, the effect of OXT varies depending on the social context and individual factors. Also, OXT-mediated effects on psychopathology and NS may depend on genetic variants of OXT receptors (OXTR). In a pilot study, the investigators demonstrated lower NS by OXT administration in a positive social context of mindfulness-based group psychotherapy (MBGT) in SSD. The investigators also demonstrated that symptoms improved after MBGT. A more recent study suggests that, compared to placebo, administering OXT in a positive social context via MBGT leads to significant between-group differences favoring OXT, particularly in NS, affect, and stress. Building on these findings, the present study investigates the stability of these effects, along with psychological and biological markers, in a larger sample of individuals with SSD. The main hypothesis to be tested is that the use of OXT compared to placebo prior to MBGT in patients with SSD will result in a greater reduction in NS with a higher OXT dosage. The research design is based on an experimental, triple-blind, randomized, placebo-controlled trial.

DETAILED DESCRIPTION:
Schizophrenia spectrum disorders (SCZ) are severe mental illnesses with a lifetime prevalence of 1-2%. Three core syndromes characterize SCZ: positive and negative syndromes (NS), as well as a cognitive syndrome. The effectiveness of current treatment options for negative symptoms (NS) and sociocognitive deficits in schizophrenia spectrum disorders (SSD) remains limited.

The cause of NS is thought to be an interference between the mesocorticolimbic dopamine system for social reward expectancy and the network for socioemotional processes. Oxytocin (OXT) may enhance functional connectivity between these neuronal networks. Lower plasma OXT levels correlate negatively with NS severity and deficits in social cognition in SSD. It has been shown that intranasal OXT administration improves social cognition in healthy subjects but in SSD results are inconsistent. According to the social salience hypothesis, the effect of OXT varies depending on the social context and individual factors. Also, OXT-mediated effects on psychopathology and NS may depend on genetic variants of OXT receptors (OXTR). In a pilot study, the investigators demonstrated lower NS by OXT administration in a positive social context of mindfulness-based group psychotherapy (MBGT) in SSD. The investigators also demonstrated that NS and other symptoms improved after MBGT. A more recent study suggests that, compared to placebo, administering OXT in a positive social context via MBGT leads to significant between-group differences favoring OXT, particularly in NS, affect, and stress. Building on these findings, the present study investigates the stability of these effects, along with psychological and biological markers, in a larger sample of individuals with SSD. The main hypothesis to be tested is that the use of OXT compared to placebo prior to MBGT in patients with SSD will result in a greater reduction in NS, i.e. the difference in T0-T8 of the total score on the BNSS (Brief Negative Symptom Scale) after 4 weeks. The BNSS as a validated rater-based instrument designed for clinical trials will be collected by a blinded psychiatrist. MBGT-sessions by experienced psychotherapists take place once a week over four weeks in a group of six patients. They serve as a positive social context for OXT administration. Participants receive either synthetic oxytocin or a placebo 30 minutes before MBGT.

The role of genetic variations (OXTR genes) for the treatment effect on NS will be explored too as well as the effect on various stress markers including cortisol levels and the endocannabinoid system, affect, group cohesion and mindfulness.

The research design is based on an experimental, triple-blind, randomized, placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Declaration of consent
* Psychiatric diagnosis of schizophrenia (ICD-10: F2x.x spectrum) for group of patients
* Mild to moderate positive symptoms (5 ≤ Positive symptoms on individual items using P-PANSS)
* German should either be the native language or spoken at a native level
* No change in systematically recorded psychopharmacological medication in the last 2 weeks before study inclusion

Exclusion Criteria:

* Acute psychotic episode with severe positive symptoms (ICD-10: F2 spectrum, 6 ≥ positive symptoms on individual items using P-PANSS)
* Acute suicidality
* Acute consumption phase of a substance dependence, except nicotine
* No severe physical impairments, neurological diseases and e.g. severe craniocerebral trauma e.g. early childhood brain damage
* Pregnancy and breastfeeding
* Current acute electroconvulsive therapy

If one of the following criteria applies to the participants, we will conduct an individual consultation in advance to determine whether participation in the study is possible:

* Overweight or underweight (body mass index (BMI) < 17.5 or > 30)
* Disease of the endocrine system
* Impaired kidney or liver function
* Metabolic diseases
* Asthma
* Change in blood potassium or sodium levels

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in BNSS Brief Negative Symptom Scale | Baseline rating (T0), post-intervention rating at week 4 (T8), follow-up 1 (week 8, T9) and follow-up 2 (week 16, T10)
  The Brief Negative Symptom Scale (BNSS) is a 13-item rater-based instrument designed for clinical trials and other studies that measures 5 domains: blunted affect, alogia, asociality, anhedonia, and avolition. The interrater, test-retest, and internal consistency of the instrument were strong, with respective intraclass correlation coefficients of 0.93 for the BNSS total score and values of 0.89-0.95 for individual subscales.

SECONDARY OUTCOMES:
Change and group differences in PANSS Negative Syndrome | Baseline rating (T0), post-intervention rating at week 4 (T8), follow-up 1 (week 8, T9) and follow-up 2 (week 16, T10)
  The Positive and Negative Syndrome Scale (PANSS) is one of the most widely used rater instruments for the assessment of the presence and severity of psychotic symptoms. Each scale comprises seven statements which are rated by the interviewer using a seven-point Likert format (from 1= absent to 7= extreme). The PANSS is reported to have satisfactory internal consistency, good interrater reliability and construct validity.
Change and group differences in SNS Self-Evaluation of Negative Symptoms | Baseline rating (T0), post-intervention rating at week 4 (T8), follow-up 1 (week 8, T9) and follow-up 2 (week 16, T10)
  The Self-Evaluation of Negative Symptoms (SNS) is a 20-item self-reported questionnaire with five subscales, namely alogia, avolition, anhedonia, social withdrawal and diminished emotional range. These subscales cluster on two factors, the apathy and emotional components. Participants can estimate the answer to each question on a scale from 0 (strongly disagree) to 3 (strongly agree). The scale was shown to have good internal consistency with Cronbach's alpha = .87.
Change and group differences in CDSS Calgary Depression Scale of Schizophrenia | Baseline rating (T0), post-intervention rating at week 4 (T8), follow-up 1 (week 8, T9) and follow-up 2 (week 16, T10)
  The Calgary Depression Scale for Schizophrenia (CDSS) is a nine item clinician rated outcome measure that assesses the level of depression in people with schizophrenia. It is the only depression scale designed to assess depression in people with a schizophrenia spectrum disorder. It distinguishes depressive symptoms from negative symptoms and is sensitive to change.
Change and group differences in PSS Perceived Stress Scale | Baseline rating (T0), post-intervention rating at week 4 (T8), follow-up 1 (week 8, T9) and follow-up 2 (week 16, T10)
  The Perceived Stress Scale (PSS) is a well-established, reliable, and valid 10-item self-report scale that measures perceived stress on a 5-point response scale (0 = "never", 1 = "almost never", 2 = "sometimes", 3 = "fairly often", 4 = "very often"). The German version of the PSS has demonstrated good internal consistency (Cronbach's α = 0.84).
Change and group differences in SMQ Southampton Mindfulness Questionnaire | Baseline rating (T0), post-intervention rating at week 4 (T8), follow-up 1 (week 8, T9) and follow-up 2 (week 16, T10)
  The Southampton Mindfulness Questionnaire (SMQ) comprises 16 items that are rated on a seven-point Likert-scale ranging from (6) "agree totally" to (0) "disagree totally". Consequently, the total score ranges from 0 to 96, with a higher score indicating higher mindfulness. The internal consistency of the German version of the SMQ was Cronbach's α = 0.89.
Change and group differences in PANAS Positive and Negative Affect Scale | Pre- and post-intervention in week 1-4 (T0-T7)
  The Positive and Negative Affect Scale (PANAS) contains 20 items, each consisting of an adjective describing an emotion. The participants have to select how applicable this adjective is to their current state from 1 (not at all) to 5 (extremely). Ten items are assigned to the positive (e.g. "Excited") as well as the negative scale (e.g. "Fearful"). The reliability of the PANAS ranges from .86 to .93.
Change and group differences in stress via visual analogue scale (Bubbles) | Pre- and post-intervention in week 1-4 (T0-T7)
  Stress via visual analogue scale. Self-rating instrument to measure stress through four items on a seven-point Likert-scale ranging from "not at all" (0) to "extreme" (6) visualized through bubbles increasing in size.
Change and group differences in GCQ-S Group Climate Questionnaire (Short Version) | Post-intervention in week 1-4 (T1, T3, T5, T7)
  The Group Climate Questionnaire [Short Version] (GCQ-S) is a 12 item questionnaire designed to assess individual group members' perceptions of the group's therapeutic environment. It consists of three domains: Engaged, conflict and avoiding and will be used as a self-report, such as a rater-based instrument.
Change and group differences in PSP Personal and Social Performance scale | Baseline rating (T0) and post-intervention rating at week 4 (T8)
  The Personal and Social Performance Scale (PSP) is a rater-based questionnaire used to assess social functioning in patients with SSD. The PSP showed good test-retest reliability (ICC = 0.79) in patients with schizophrenia.
Change and group differences in endocannabinoid levels | Pre- and post-intervention in week 1 (T0, T1), post-intervention in week 4 (T7) and follow-up 1 (week 8, T9)
  Venous blood samples will be taken to determine the endocannabinoid levels to obtain an individual baseline and comparison level.
Change and group differences in interleukin levels | Pre-intervention in week 1 (T0) and post-intervention in week 4 (T7)
  Venous blood samples will be taken to determine the interleukin levels to obtain an individual baseline and comparison level.
Change and group differences in oxytocin levels | Pre- and post-intervention in week 1 (T0, T1) and post-intervention in week 4 (T7)
  Venous blood samples will be taken to determine the oxytocin levels to obtain an individual baseline and comparison level.
Change and group differences in PBMC levels | Pre-intervention in week 1 (T0) and post-intervention in week 4 (T7)
  Venous blood samples will be taken to determine the PBMC levels to obtain an individual baseline and comparison level.
Change and group differences in cortisol saliva levels | Pre- and post-intervention in week 1-4 (T0-T7)
  Saliva samples will be taken before and after each MBGT session to determine Cortisol saliva levels

CONTACTS AND LOCATIONS:
Overall Officials: Marco Zierhut, MD, Principal Investigator — Charite University, Berlin, Germany; Kerem Böge, Prof., Principal Investigator — Charite University, Berlin, Germany; Eric Hahn, PD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin, Campus Benjamin Franklin, Campus Charité Mitte, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boge K, Bergmann N, Zierhut M, Hahne I, Braun A, Kraft J, Conell I, Ta TMT, Thomas N, Chadwick P, Ripke S, Hahn E. The relationship between mindfulness and empathy with the oxytocinergic system in persons with schizophrenia spectrum disorders - A proof-of-concept randomized controlled trial (OXYGEN). Int J Clin Health Psychol. 2024 Jul-Sep;24(3):100503. doi: 10.1016/j.ijchp.2024.100503. Epub 2024 Sep 10. PMID 39308779
- [Background] Zierhut M, Bergmann N, Hahne I, Wohlthan J, Kraft J, Braun A, Tam Ta TM, Hellmann-Regen J, Ripke S, Bajbouj M, Hahn E, Boge K. The combination of oxytocin and mindfulness-based group therapy for empathy and negative symptoms in schizophrenia spectrum disorders - A double-blinded, randomized, placebo-controlled pilot study. J Psychiatr Res. 2024 Mar;171:222-229. doi: 10.1016/j.jpsychires.2024.01.014. Epub 2024 Jan 9. PMID 38309212
- [Background] Boge K, Hahne I, Bergmann N, Wingenfeld K, Zierhut M, Thomas N, Ta TMT, Bajbouj M, Hahn E. Mindfulness-based group therapy for in-patients with schizophrenia spectrum disorders - Feasibility, acceptability, and preliminary outcomes of a rater-blinded randomized controlled trial. Schizophr Res. 2021 Feb;228:134-144. doi: 10.1016/j.schres.2020.12.008. Epub 2021 Jan 9. PMID 33434727